CLINICAL TRIAL: NCT00981461
Title: A Randomized, Double-Blind Clinical Trial to Evaluate the Safety and Efficacy of the HairMax LaserComb 2009, 9 Beam Model: For the Treatment of Androgenetic Alopecia in Females
Brief Title: Treatment of Androgenetic Alopecia in Females, 9 Beam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lexington International, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 151.0805
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Androgenetic Alopecia; Hair Loss; Female Pattern Baldness
Keywords: Andregenetic Alopecia; Hair Loss; Female Pattern Baldness
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLT Device 2009 9 Beam (Active Comparator): HairMax LaserComb
  Interventions: Device: HairMax LaserComb
- control device (Sham Comparator): control device
  Interventions: Device: Control Device

INTERVENTIONS:
Device: HairMax LaserComb — Device application 3 times week, for 26 weeks
  Arms: LLT Device 2009 9 Beam
Device: Control Device — Device application 3 times week, for 26 weeks
  Arms: control device

SUMMARY:
The purpose of this study is to evaluate the efficacy of the HairMax LaserComb 2009 9 beam model in promoting hair growth in females diagnosed with androgenetic alopecia when treatment is applied as directed.

DETAILED DESCRIPTION:
This is a randomized double-blind, control device clinical study across 5 sites, evaluating changes in terminal hair count in the evaluation zone having evidence of androgenetic alopecia (miniaturized hair).

The trial with 60 female subjects who have been diagnosed with androgenetic alopecia, who are between 25 and 60 years of age, have Fitzpatrick Skin Types I-IV, with classifications of Ludwig I-4, II-1, II-2, or frontal, have active hair loss within the last 12 months.

Subjects will use the device on three non-concurring days a week as directed per device for 26 weeks duration.

Initial efficacy endpoint for each subject will be assess at visit 4 (week 16).

Safety analysis will be assessed based on the reports of adverse events during study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of androgenetic alopecia
* Fitzpatrick Skin Types I-IV
* Ludwig I-4, II-1, II-2, or frontal
* Active hair loss within last 12 months

Exclusion Criteria:

* Photosensitivity to laser light
* Malignancy in the target area
* Pregnancy
* Lactating females

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jarratt, M.D., Principal Investigator — DermaResearch, Inc.; Abe Marcadis, M.D., Principal Investigator — Palm Beach Research Center; David Goldberg, M.D., Principal Investigator — Hackensack, NJ; Neil S Sadick, MD, Principal Investigator — Sadick Research Group; Jose Mendez, DO, Principal Investigator — International Dermatology Research, Inc.; Janet Hickman, MD, Principal Investigator — The Education and Researvh Foundation
Locations (5):
- United States (5):
  - Jose Mendez, DO, Miami, Florida
  - Abe Marcadis, MD, Palm Beach, Florida
  - David Goldberg, MD, Hackensack, New Jersey
  - Sadick Research Group, New York, New York
  - Janet Hickman, MD, Lynchburg, Virginia

REFERENCES:
- [Result] Leavitt M, Charles G, Heyman E, Michaels D. HairMax LaserComb laser phototherapy device in the treatment of male androgenetic alopecia: A randomized, double-blind, sham device-controlled, multicentre trial. Clin Drug Investig. 2009;29(5):283-92. doi: 10.2165/00044011-200929050-00001. PMID 19366270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind, device controlled 26 week study was recruited at 6 clinical study sites. The recruitment period was from October 29, 2008 to March 2, 2009
Pre-assignment Details: Key exclusion criteria was pregnancy, malignancy in target area, an no hair transplants, scalp reductions, or hair weaves. Active hair loss less than 12 months.
Groups:
- HairMax LaserComb 2009 9 Beam: This arm involves the active LLLT device with 9 laser modules. The device is used 3 times a week for 12 minutes per session for full 26 duration of the study. This device was distributed to subjects in a blinded randomized manner. Subjects were evaluated at 8, 16 and 26 weeks, with hair counts performed at week 16 and 26.
- Control Device: This arm involves the use of an inactive control device that emits white light. The device is used 3 times a week for full 26 duration of study. This arm of the study was blinded and dispensed to subjects on a random basis.Subjects were evaluated at 8, 16 and 26 weeks, with hair counts performed at week 16 and 26.
Period: Overall Study
Arm/Group | HairMax LaserComb 2009 9 Beam | Control Device
Started | 48 | 24
Completed | 43 | 22
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- HairMax LaserComb 2009 9 Beam: This arm involves the active LLLT device with 9 laser modules. The device is used 3 times a week for 12 minutes per session for full length of study. This device was distributed to subjects in a blinded randomized manner
- Control Device: This arm involves the use of an inactive control device that emits white light. The device is used 3 times a week for full length of study. This arm of the study was blinded and dispensed to subjects on a random basis.
- Total: Total of all reporting groups
Arm/Group | HairMax LaserComb 2009 9 Beam | Control Device | Total
Number analyzed (Participants) | 43 | 22 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 22 | 65
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 22 | 65
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Terminal Hair Count Week 16 and 26 Weeks Over Baseline
Description: The primary analysis of effectiveness was an analysis of covariance, which separately modeled terminal hair count at Week 16 and Week 26 as a function of treatment group (HairMax LaserComb 2009 9 Beam vs.control), study center, age (as a continuous variable), and Fitzpatrick Skin Type classification (as a categorical variable with four levels). The active group was compared to the control device using least squares means with a two-sided test at the 5% level of significance.
Time Frame: Baseline, 16 weeks, 26 weeks
Measure: Mean (Standard Deviation); unit: hairs per cm^2
Groups:
- Control Device: This control device is inactive emitting white light
- HairMax LaserComb 2009 9 Beam: This device is the active device with 9 laser modules
Arm/Group | Control Device | HairMax LaserComb 2009 9 Beam
Number analyzed (Participants) | 22 | 43
hairs per cm^2
  Change at 16 weeks | 1.3 (14.67) | 14.8 (9.70)
  Change at 26 weeks | 2.8 (16.48) | 20.2 (11.15)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Device | HairMax LaserComb 2009 9 Beam
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/43
Other Adverse Events (participants affected / at risk) | 0/22 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No